CLINICAL TRIAL: NCT01611753
Title: Red Blood Cell Transfusion Improves Perfusion Parameters in Septic Shock Patients With Hypoperfusion: a Prospective Randomized Study
Brief Title: Red Blood Cell Transfusion Improves Perfusion Parameters in Septic Shock Patients With Hypoperfusion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bruno Franco Mazza (Other)
Responsible Party: Sponsor-Investigator, Bruno Franco Mazza, MD, Federal University of São Paulo
Organization: Federal University of São Paulo (Other)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 1177/04
Record Dates: First submitted 2012-05-24; First posted 2012-06-05 (Estimated); Last update posted 2012-06-05 (Estimated); Status verified 2012-05

CONDITIONS: Septic Shock
Keywords: Shock, Septic; Erythrocyte Transfusion; Ischemia
MeSH Terms: conditions — Shock, Septic; Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- liberal group (Active Comparator): Patients in the liberal group received transfusions immediately, as the objective was to maintain hemoglobin levels above 9.0 g/dL.
  Interventions: Other: packed red blood cell transfusion
- restrictive group (Active Comparator): Patients in the liberal group received transfusions immediately, as the objective was to maintain hemoglobin levels above 7.0 g/dL.
  Interventions: Other: packed red blood cell transfusion

INTERVENTIONS:
Other: packed red blood cell transfusion — Patients wil be randomized en two groups, in the liberal group they must received transfusions immediately, as the objective was to maintain hemoglobin levels above 9.0 g/dL. In the restrictive group they will receive transfusion to maintain hemoglobin levels above 7.0g/dL

SUMMARY:
The purpose of this study was to evaluate the immediate effects of red blood cells transfusion on central venous oxygen saturation and lactate levels in septic shock patients randomized to two different hemoglobin levels.

The influence of red blood cell (RBC) transfusion on the adequacy of oxygen delivery (DO2) and supply (VO2) could be assessed by systemic oxygen variables such as central venous oxygen saturation (ScvO2) and lactate levels. Although it is not clear that alterations in these parameters actually represent an improvement in the DO2/VO2 ratio, they might represent a better transfusion trigger than the absolute hemoglobin value.

Patients admitted with a diagnosis of septic shock and hemoglobin levels lower than 9.0 g/dL , less than 48 hours of shock diagnosis, were included, a central venous catheter in the superior vena cava and signed informed consent. The investigators randomized all patients into two groups. Patients in the liberal group received transfusions immediately, as the objective was to maintain hemoglobin levels above 9.0 g/dL. In the restrictive group, transfusion was withheld until their hemoglobin levels fell below 7.0 g/dL.

Each time a patient received a transfusion, the investigators collected a set of laboratory tests, including hemoglobin levels, ScvO2 and lactate, at two time points, immediately before transfusion and one hour after its ending.

The sample size was calculated by considering that in 80% of the transfusions in patients in the restrictive group ScvO2 would improve compared to only 45% of those in the liberal group, with an alpha error of 0.05 and 80% power. Improvement was defined as an increase of 5% over the pre-transfusion ScvO2. Twenty-eight transfusions in each group would be necessary, but to correct for potential non-parametric distribution of the main variables, the number was adjusted to 35 transfusions in each group.

Trends in ScvO2 and lactate were categorized as worsening or improving. The investigators defined improvement when ScvO2 reached 70% in patients with baseline levels below this threshold or when there was an absolute increase of at least 5% after transfusion. Any increase in patients with previous ScvO2 ≥ 70% was considered to be "no change". Worsening was defined as a reduction of 5% in the previous levels or a decline to less than 70% in patients with pre-transfusion levels in the range of 70 to 75%. The investigators also carried out a ROC curve analysis to assess the accuracy of the pre-transfusion hemoglobin levels, pre-transfusion lactate and pre-transfusion ScvO2 in predicting the patients whose ScvO2 would increase more than 5% with transfusion. For this analysis, the investigators used a different approach because it would also be necessary to analyze patients with a lower chance of response to assess the prediction of response. Thus, this analysis included all patients with ScvO2 below 75%, rather than only those below 70%. As before, the investigators defined improvement as any increase ≥ 5%. The investigators did not consider patients with levels above 75% in this analysis, as the physiological interpretation of this situation is challenging. The investigators considered as altered any lactate levels above 1.5 times the reference level, and a change ≥ 10% was defined as improvement or worsening. In patients with baseline normal levels, the status was recorded as worsening if a 10% increase was detected. Afterwards, the investigators tested the association between these categorized variables and the baseline levels of hemoglobin. The impact on perfusion was also assessed by the determination of Δlactate (lactate post-transfusion x 100/lactate pre-transfusion) and ΔScvO2 (ScvO2 post-transfusion x 100/ScvO2 pre-transfusion), and their correlation with the baseline hemoglobin levels was analyzed using the Spearman correlation test.

In all tests, the results were considered significant if the p level was lower than 0.05.

ELIGIBILITY:
Inclusion Criteria:

* age over 18 years old
* less than 48 hours of shock diagnosis
* hemoglobin levels lower than 9.0 g/dL
* a central venous catheter in the superior vena cava
* signed informed consent. The exclusion criteria were

Exclusion Criteria:

* pregnancy
* known coronary disease
* active bleeding
* previous participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2004-04; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Evaluate the change in baseline levels of lactate and central venous saturation effects after red blood cells transfusion in patients of septic shock | The purpose of this study was to evaluate the effects of red blood cells transfusion on central venous oxygen saturation and lactate levels after 1 hour in septic shock patients randomized to two different hemoglobin levels

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Sao Paulo - Universitary hospital of Sao Paulo Federal University, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Mazza BF, Freitas FG, Barros MM, Azevedo LC, Machado FR. Blood transfusions in septic shock: is 7.0 g/dL really the appropriate threshold? Rev Bras Ter Intensiva. 2015 Jan-Mar;27(1):36-43. doi: 10.5935/0103-507X.20150007. Epub 2015 Mar 1. PMID 25909311